CLINICAL TRIAL: NCT01316003
Title: Distinction of Cone Outer Segment Tips by Spectral-Domain Optical Coherence Tomography in Normal Eyes
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor, Kyorin University
Other Study IDs: KyorinEye004
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: cone outer segment tips line; Optical coherence tomography
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal subjects: Thirty-seven eyes of 37 individuals without eye diseases
  Interventions: Other: Optical coherence tomography

INTERVENTIONS:
Other: Optical coherence tomography — Optical coherence tomography
  Other Names: Cirrus HD-OCT (Carl Zeiss Meditec)

SUMMARY:
The aim of this study is to investigate the incidence and possible causes of obscured or disrupted cone outer segment tips line at fovea in spectral-domain optical coherence tomography images of normal eyes.

DETAILED DESCRIPTION:
Thirty-seven eyes of 37 individuals without eye diseases were included in this study. Optical Coherence Tomography (OCT) images were taken using Cirrus HD-OCT (Carl Zeiss Meditec) with 5 line raster and high-definition 5 line raster modes. Images with signal strength weaker than 5/10 were excluded. Distinction of COST line and the integrity of COST line, external limiting membrane, and the photoreceptor inner segment and outer segment junction at the fovea were recorded. Demographic data, refractive error of the eyes, signal strengths of the OCT images were acquired for analysis.

ELIGIBILITY:
Inclusion Criteria:

* individuals without eye diseases

Exclusion Criteria:

* individuals with eye diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty-seven eyes of 37 individuals without eye diseases
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Microstructural analysis by Spectral domain optical coherence tomography | one year
  SD-OCT images of 6 mm scans were taken using Cirrus HD-OCT (OCT 4000, Carl Zeiss Meditec, Dublin, CA) with 5 line raster (5LR) and high-definition 5 line raster (HD5LR) modes.

SECONDARY OUTCOMES:
Visual acuity | one year
  Each subject had a routine eye examination including measuring best-corrected visual acuity (BCVA) and intraocular pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan

REFERENCES:
- [Derived] Rii T, Itoh Y, Inoue M, Hirakata A. Foveal cone outer segment tips line and disruption artifacts in spectral-domain optical coherence tomographic images of normal eyes. Am J Ophthalmol. 2012 Mar;153(3):524-529.e1. doi: 10.1016/j.ajo.2011.08.021. Epub 2011 Oct 21. PMID 22018706